CLINICAL TRIAL: NCT06882967
Title: Thoracic Endovascular Aortic Repair in Compromised Distal Landing Zones
Brief Title: Active Thoracic Compromised Distal LANding in TEvar
Acronym: ATLANTE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5107
Record Dates: First submitted 2023-03-09; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Aortic Aneurysm; Aortic Diseases
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Diseases | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Distal active fixation stent-grafts: Distal active fixation stent-grafts
  Interventions: Device: Thoracic Endovascular Aortic Repair
- Distal scallop stent-grafts: Distal scallop custom-made stent-grafts
  Interventions: Device: Thoracic Endovascular Aortic Repair
- Distal Aptus Heli-FX EndoAnchors: Distal Aptus Heli-FX EndoAnchors
  Interventions: Device: Thoracic Endovascular Aortic Repair
- Standard stent-grafts: Standard Thoracic stent-graft
  Interventions: Device: Thoracic Endovascular Aortic Repair

INTERVENTIONS:
Device: Thoracic Endovascular Aortic Repair — Placement of a covered stent (a metal mesh tube with a layer of fabric) into the weakened area of the artery.

SUMMARY:
Thoracic endovascular aortic repair (TEVAR) has become the mainstay of aortic intervention for descending thoracic aortic pathology. Its durability hinges on achieving adequate seal in the endograft landing zones (LZs), with the distal LZ largely understudied. Only recently are suboptimal distal LZs receiving attention for their role in major complications including stent graft migration, type 1B endoleaks, and distal stent graft-induced new entry tears, all of which can contribute to further aortic degeneration. The thoracic distal LZ. When a short distal LZ was reported, the distal endoleak rate ranged from 3.5% to 33%. This led to reintervention in 19%, along with coverage of the celiac trunk in more than half of short LZ cases.

The objective of this study was to evaluate the outcomes of TEVAR patients with compromised distal landing zone (CDLZs) treated with distal active fixation stent-grafts (DAFs), distal scallop stent-grafts, distal Aptus Heli-FX EndoAnchors, and standard stent-grafts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with descending thoracic aortic aneurysms (DTAAs) with a maximal aortic diameter > 55mm or rapid growth (>10mm / year).
* Patients presenting with at least 2 cognizable features related to an adverse aortic morphology will be considered for inclusion. The following features will be evaluated for the inclusion: distal LZ length ≤25-mm, distal LZ diameter ≥38-mm, LZ conical morphology, distal descending thoracic aorta angulation ≤116° or tortuosity index ≥1.4

Exclusion Criteria:

* Emergency setting, including hemodynamic instability at time of enrollment
* Patients with aortic dissection pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with compromised distal landing zone undergoing Thoracic Endovascular Aortic Repair in patients with distal active fixation stent-grafts, distal scallop stent-grafts, distal EndoAnchors, and standard stent-grafts in selected high volume aortic centers will be enrolled retrospectively with a prospective database
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Ib Endoleak | Follow-up (at month 3)
  Presence of type Ib endoleak

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No